CLINICAL TRIAL: NCT00838058
Title: An Open-Label Two-Part Randomized, Crossover Study Of The Pharmacokinetics Of CE-224,535 Administered As Controlled And Immediate Release Formulations In Healthy Volunteers
Brief Title: A Study in Normal Healthy People, Testing Different Versions of a Pill That Will be Used to Treat Rheumatoid Arthritis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A6341012
Record Dates: First submitted 2009-02-02; First posted 2009-02-06 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Rheumatoid Arthritis; Healthy Volunteers
Keywords: pharmacology formulation normal healthy volunteers food effect
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CE 224,535

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part1; controlled release formulation 4; 250 mg (Experimental): one 250 mg controlled release tablet, once in the morning, in fasted state
  Interventions: Drug: CE-224,535
- Part1; controlled release formulation 4; 500 mg (Experimental): 2x250 mg, once in the morning, in fasted state
  Interventions: Drug: CE-224,535
- Part 1; controlled release formula 4; 1000 mg (Experimental): 4x250 mg tabs, once in the morning, in fasted state
  Interventions: Drug: CE-224,535
- Part 1; controlled release formulation 4; 500 mg FED (Experimental): 2x250 mg, once in the morning , in fed state
  Interventions: Drug: CE-224,535
- Part 2; IR formulation 500mg (Experimental): 4x125 mg tab of current formulation , once in the morning in the fasted state. This arm will occur as Part 2, only as needed, pending results of Part 1
  Interventions: Drug: CE-224,535
- Part 2; IR formulation, 500 mg FED (Experimental): 4x125 mg once in the morning in the fed state. This arm will occur as part of Part 2,only as needed, pending results of Part 1.
  Interventions: Drug: CE-224,535
- Part 2; controlled release formulation 5;500 mg, FASTED (Experimental): 2x250 controlled release formulation 5 tabs once in the morning in the fasted state. This arm will only occur as part of Part 2, pending results of Part 1.
  Interventions: Drug: CE 224,535
- Part 2; controlled release formulation 5;500 mg, FED (Experimental): 2x250 mg controlled release formulation 5 tabs once in the morning in the fed state. This arm will only occur as part of Part 2 pending results of Part 1
  Interventions: Drug: CE 224,535

INTERVENTIONS:
Drug: CE-224,535 — one 250mg tablet, once in the morning in fasted state
  Other Names: Part 1;Treatment A
  Arms: Part1; controlled release formulation 4; 250 mg
Drug: CE-224,535 — 2x250 mg tablets, once in the morning, in fasted state
  Other Names: Part 1;Treatment B
  Arms: Part1; controlled release formulation 4; 500 mg
Drug: CE-224,535 — 4x250mg tablets, once in the morning, in fasted state
  Other Names: Part 1;Treatment C
  Arms: Part 1; controlled release formula 4; 1000 mg
Drug: CE-224,535 — 2x250mg tab, once in the morning, after being fed a high fat meal
  Other Names: Part 1;Treatment D
  Arms: Part 1; controlled release formulation 4; 500 mg FED
Drug: CE-224,535 — 4x125 mg tabs, once in the morning, in the fasted state. This arm will only occur as part of Part 2, if needed, pending results of Part 1.
  Other Names: Part 2;Treatment E
  Arms: Part 2; IR formulation 500mg
Drug: CE-224,535 — 4x125 mg IR once in the morning after being fed a high fat meal
  Other Names: Part 2; Treatment F
  Arms: Part 2; IR formulation, 500 mg FED
Drug: CE 224,535 — 2x250 mg controlled release formulation 5 tabs once in the morning in the fasted state
  Other Names: Part 2; Treatment G
  Arms: Part 2; controlled release formulation 5;500 mg, FASTED
Drug: CE 224,535 — 2x250 mg controlled release formulation 5 once in the morning after being fed a high fat meal
  Other Names: Part 2; Treatment H
  Arms: Part 2; controlled release formulation 5;500 mg, FED

SUMMARY:
The study will try, in 2 separate parts, each using 12 research subjects, to see how a new form of the pill CE 224,535 gets released into the bloodstream and whether that is affected by food. In each part, subjects will switch among 4 treatment periods to take either different forms of the pill(s) or the same form either after fasting or eating a meal. The second part will only happen depending on whether the sponsor believes it is needed and will use separate subject than the first part.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-55 and healthy

Exclusion Criteria:

* severe chronic or uncontrolled medical or psychiatric conditions, including drug abuse
* pregnant or wanting to become pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters: Tmax, Cmax, AUClast, AUC(0-00), C24, t1/2 | 48 hrs

SECONDARY OUTCOMES:
safety parameters including: renal and liver function, blood counts, electrolytes, ECG, and pregnancy testing | 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6341012&StudyName=A%20study%20in%20normal%20healthy%20people%2C%20testing%20different%20versions%20of%20a%20pill%20that%20will%20be%20used%20to%20treat%20rheumatoid%20arthritis.